CLINICAL TRIAL: NCT06742307
Title: Faricimab Fixed Quarterly Maintenance for Neovascular Age Related Macular Degeneration: A Prospective Case Series
Brief Title: Faricimab Quarterly Maintenance for Neovascular Age Related Macular Degeneration
Acronym: Fixed farcimab
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Authority, Hong Kong (Other Government)
Responsible Party: Principal Investigator, Wong Ho Daniel Tak, Principal Investigator, Hospital Authority, Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIRB-2024-169-3
Record Dates: First submitted 2024-12-15; First posted 2024-12-19 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Macular Degeneration Choroidal Neovascularization
Keywords: neovascular age related macular degeneration; faricimab
MeSH Terms: conditions — Choroidal Neovascularization | interventions — faricimab

STUDY DESIGN:
Intervention Model Description: Patients included, once diagnosed with neovascular macular dengeration, will embark on a planned quarterly (every 12-16 weeks) faricimab injection schedule for one year, following a disease inactivity achieved after initial 2-4 loading doses of faricimab. If disease inactivity is not achieved during the maintenance phase, patient's injection interval may be shortened.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Faricimab treatment arm (Active Comparator): A planned quarterly (every 12-16 weeks) faricimab injection schedule, following a disease inactivity achieved after initial 2-4 loading doses of faricimab. The intervention faricimab is injected into the eyeball with a 30G needle.
  Interventions: Drug: Faricimab Injection [Vabysmo]

INTERVENTIONS:
Drug: Faricimab Injection [Vabysmo] — A planned quarterly (every 12-16 weeks) faricimab injection schedule, following a disease inactivity achieved after initial 2-4 loading doses of faricimab. This intervention schedule is not specifically studied in other literature, although similar schedule exist.

SUMMARY:
We aimed to investigate the success rate of a planned quarterly (every 12-16 weeks) faricimab injection schedule, following a disease inactivity achieved after initial 2-4 loading doses of faricimab, for nAMD to achieve stability without recurrence at a tertiary eye centre.

DETAILED DESCRIPTION:
Age-related macular degeneration (AMD) accounts for 8.7% of all causes of blindness worldwide and is the most common cause of blindness in developed nations. Its prevalence is likely to increase as a consequence of exponential population ageing. Wet, or neovascular, AMD affects 10-15% of AMD patients and is characterised by macular neovascularisation (MNV), where new immature blood vessels grow towards the outer retina, typically from the underlying choroid, result in leakage, fluid accumulation, and haemorrhage. Faricimab is a bispecific antibody that acts through dual inhibition of both angiopoietin-2 and vascular endothelial growth factor A (VEGF-A). Safety and efficacy of intravitreal faricimab were evaluated in phase 3 trials in patients with nAMD. TENAYA and LUCERNE assessed faricimab administered at individualised treatment intervals of up to every 16 weeks compared with aflibercept given every 8 weeks in patients with nAMD.

Different treatment regimens exist, including the pro re nata (PRN) and the treat and extend (T&E) approaches. Treating macular disease with anti-VEGF has been an enormous burden to ophthalmic services globally. In Hong Kong, anti-VEGF treatment is self-financed, hindering access for the underprivileged. It has been mentioned that most public hospitals in the region are less likely to adopt a T&E regimen directly after the loading phase but are more inclined towards PRN regimen because of limited manpower and resources .

Generally, three monthly or four-weekly anti-VEGF injections before the introduction of faricimab to the public hospitals in Hospital Authority (HA) in 2023 would be arranged for newly diagnosed patients with nAMD during the initial visit at our institution. Depending on the treatment response, the patient would either be advised to stop injections (PRN regimen), to T&E regimen by extending the intervals in a stepwise manner, or be put on regular quarterly maintenance injections.

From the full prescribing information supplied by the manufacturer Roche, for nAMD, the recommended dose for Vabysmo® (Faricimab) is 6 mg (0.05 mL of 120 mg/mL solution) administered by intravitreal injection every 4 weeks (approximately every 28 ± 7 days, monthly) for the first 4 doses (at Weeks 0, 4, 8, 12), followed by optical coherence tomography (OCT) and visual acuity evaluations 8 and 12 weeks later to inform whether to give a 6 mg dose via intravitreal injection on one of the following three regimens: 1) Weeks 28 and 44 (every 16 weeks); 2) Weeks 24, 36 and 48 (every 12 weeks); or 3) Weeks 20, 28, 36 and 44 (every 8 weeks). Although additional efficacy was not demonstrated in most patients when Vabysmo® was dosed every 4 weeks compared to every 8 weeks, some patients may need every 4 week (monthly) dosing after the first 4 doses. Patients should be assessed regularly.

As this new drug, faricimab, is becoming available in the hospital authority (HA) in Hong Kong, it is expected to be more extensively given to our patients with nAMD. It is understood from the full prescribing information supplied by Roche that the injection interval can be extended up to 16 weeks. It is vital to have the knowledge whether some less treatment intensive, simple fixed regimen in our locality is comparable to the more intensive dosing suggested by the manufacturer. With the number of injections administered in the territory exponentially rising in recent years due to the ageing population, there is clearly a need to explore better alternatives to the PRN approach and this forms the basis of our study.

ELIGIBILITY:
Inclusion Criteria:

Subjects aged over 50 years, neovascular AMD with foveal involvement, both treatment-naïve and recurrent cases. There were no specific criteria for initial best-corrected visual acuity (BCVA). Only active subfoveal MNV are included, including types 1, 2, and 3.

Exclusion Criteria:

* eyes that received any anti-VEGF therapy in the prior six months,
* eyes with other disease entities (e.g., diabetic macula oedema, retinal vein occlusions, central serous chorioretinopathy, myopicmacular neovascularisation),
* concurrent macula laser (except photodynamic therapy) and ocular surgery (e.g., cataract surgery or vitrectomy) in the prior six months and the study period.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-08-21 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Visual acuity | 52 weeks
  The primary outcome is the change from baseline in best-corrected visual acuity (BCVA) at week 52.

SECONDARY OUTCOMES:
Anatomical success | 52 weeks
  Anatomical success was defined as no increase in disease activity of the AMD on clinical examination or OCT throughout the study period while remaining on the quarterly dosing schedule, without the need to shorten the treatment interval.
Functional success | 52 weeks
  Functional success was characterised by a loss of fewer than five ETDRS letters, without the need to shorten the treatment interval.
Maintenance treatment failure | 52 weeks
  Maintenance treatment failure was defined as an increase in disease activity during the quarterly dosing maintenance stage, i.e. new macular haemorrhage, neovascularisation, and/or an increase in OCT biomarkers for neovascular activity, and thus a decision for rescue treatment with shorter treatment intervals.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Ophthalmology, United Chrisitian Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Patient number and enrollment status.
Supporting Information: Study Protocol
Time Frame: 6/2025 for 2 years till 6/2027
Access Criteria: Other researches submitting such request to us. they will be able to access the research protocol and current enrollment status. No patient information will be shared. They can access it by sending us the request. We will seek advice from our local ethics committee CIRB for advice for entertaining such requests.

REFERENCES:
- [Background] Wong DHT, Li KKW. Fixed Quarterly Dosing of Aflibercept after Loading Doses in Neovascular Age-Related Macular Degeneration in Chinese Eyes. J Clin Med. 2023 Dec 27;13(1):145. doi: 10.3390/jcm13010145. PMID 38202151
- [Background] Heier JS, Khanani AM, Quezada Ruiz C, Basu K, Ferrone PJ, Brittain C, Figueroa MS, Lin H, Holz FG, Patel V, Lai TYY, Silverman D, Regillo C, Swaminathan B, Viola F, Cheung CMG, Wong TY; TENAYA and LUCERNE Investigators. Efficacy, durability, and safety of intravitreal faricimab up to every 16 weeks for neovascular age-related macular degeneration (TENAYA and LUCERNE): two randomised, double-masked, phase 3, non-inferiority trials. Lancet. 2022 Feb 19;399(10326):729-740. doi: 10.1016/S0140-6736(22)00010-1. Epub 2022 Jan 24. PMID 35085502
- [Background] Wong WL, Su X, Li X, Cheung CM, Klein R, Cheng CY, Wong TY. Global prevalence of age-related macular degeneration and disease burden projection for 2020 and 2040: a systematic review and meta-analysis. Lancet Glob Health. 2014 Feb;2(2):e106-16. doi: 10.1016/S2214-109X(13)70145-1. Epub 2014 Jan 3. PMID 25104651
- [Background] Ambati J, Fowler BJ. Mechanisms of age-related macular degeneration. Neuron. 2012 Jul 12;75(1):26-39. doi: 10.1016/j.neuron.2012.06.018. PMID 22794258
- See also: Genentech, Inc, Roche Group. HIGHLIGHTS OF PRESCRIBING INFORMATION. — https://www.gene.com/download/pdf/vabysmo_prescribing.pdf